CLINICAL TRIAL: NCT04835909
Title: Effectiveness on Cognition of a Cognitive Training Intervention Based on Modern Board and Card Games in Mild Cognitive Impairment Patients: a Randomized Controlled Trial
Brief Title: Board Games Among Mild Cognitive Impairment Patients Experience (GAME Project)
Acronym: GAME-Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brain In Game scientific-technical service (Other)
Collaborators: University Hospital of Santa Maria, Lleida (Unknown)
Responsible Party: Principal Investigator, jaume march llanes, Effectiveness on Cognition of a Cognitive Training Intervention Based on Modern Board and Card Games in Mild Cognitive Impairment Patients: a Randomized Controlled Trial, Brain In Game scientific-technical service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCT2021UTC
Record Dates: First submitted 2021-03-22; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Impairment, Mild
Keywords: Memory; Executive Functions; Cognitive training; Cognitive enrichment; Modern board and card games
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Paper

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral: modern board and card games (Experimental): Participants will play modern board and card games in groups at medical center 2 times per week for at least 1 hour over a period of 16 weeks.
  Interventions: Behavioral: Modern board and card games group
- Behavioral: paper and pencil tasks (Active Comparator): Participants will do cognitive paper and pencil tasks in groups at medical center 2 times per week for at least 1 hour over a period of 16 weeks.
  Interventions: Behavioral: Paper and pencil tasks group
- Wait-list (No Intervention): Participants will be in a wait-list over a period of 16 weeks. Then, they received the board and card games' or paper and pencil tasks' intervention.

INTERVENTIONS:
Behavioral: Modern board and card games group — Modern board and card games group
  Arms: Behavioral: modern board and card games
Behavioral: Paper and pencil tasks group — Paper and pencil tasks group
  Arms: Behavioral: paper and pencil tasks

SUMMARY:
Nowadays, on geriatric centres, cognitive decline used to be prevented by pen and paper exercises (Calero García & Navarro Gonzalez, 2006). However, as Lampit et al. (2014) suggest, studies based on the efficacy and effectiveness of new cognitive-based interventions in order to improve these cognitive processes are fundamental (Lampit et al., 2014). Cognitive-based interventions are interventions that directly or indirectly try to improve cognitive processes (Chiu et al., 2017). Between the different kinds of cognitive-based interventions, cognitive training permits stablish randomized controlled trials. Cognitive training consists of repeating during a concrete time a standardized set of tasks in order to maintain or improve one or some cognitive processes. Meta-analysis studies have shown that computerized cognitive training can improve in a moderate size some cognitive processes in elderly people with mild cognitive impairment or dementia (Hill et al., 2017) and without those diagnoses (Lampit, Hallock, & Valenzuela, 2014; Chiu et al., 2017). Although it seems that computerized training is effective, safe and secure, it is important to note the social component of the definition of health (OMS, 1948). Chang, Wray & Lin (2014) found that social relationships predict the use of leisure activities and this predict a better physical health and wellbeing psychological. In fact, a comparative study found that those elderly people that have played board games have a 15% lower risk of having dementia diagnose and problems related with memory (Dartigues et al., 2013). To sum up, the aim of this research project is to test the effectiveness of a cognitive training based on modern board and card games in elderly people with a diagnose of mild-cognitive impairment in comparison to do cognitive paper and pencil tasks or in a wait-list comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Participation in cognitive disease center
* Amnestic MCI diagnoses (clinical diagnoses following the guidelines of Petersen et al. 2011)
* Global deterioration scale (GDS) 2-3 values
* Participation assessing outcomes of the caregivers in the study

Exclusion Criteria:

* Participation in another cognitive training program
* Dementia, neurologic or other disease non-neurodegenerative, which could affect cognitive change over time (medical-reported)
* Severe visual impairment, language impairment or motoric impairment of the upper extremity which significantly affects ability to solve jigsaw puzzles (medical-reported)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive impairment from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Addenbrooke's Cognitive Examination
Change in visuoconstruction, immediate memory and long-term memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Copy, draw after 3 and after 25 minuts of Rey-Osterrieth Complex Figure Test
Change in verbal long-term memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Rey Auditory Verbal Learning Test (RAVLT)
Change in verbal short-term memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Digit Memory Test Forward
Change in verbal working memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Digit Memory Test Backward
Change in visuospatial short-term memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Visual Memory Test Forward
Change in visuospatial working memory from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Visual Memory Test Backward
Change in visuospatial processing from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Trail Making Test A and Symbol Digit Modalities Test (SDMT)
Change in flexibility from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Trail Making Test B and 5 digits test
Change in inhibition from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  5 digits test
Change in phonemic and semantic fluency from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Animals category and P, M, R letters, Spanish version

SECONDARY OUTCOMES:
Change in neuropsychiatric symptoms from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Neuropsychiatric Inventory (NPI), Self-reported and caregivers spanish versions. Higher scores mean higher neuropsychiatric symptomatology.
Change in psychological well-being from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Euro Quality of Life Scale (EQ-5D), Self-reported and caregivers spanish versions. Higher scores mean higher quality of life. Visual analogue scale: minimum value=0, maximum value=100.
Change in depressive symptoms from baseline to post intervention | Baseline and post intervention (after 16 weeks)
  Geriatric Depression Scale (GDS), Spanish version. Higher scores mean higher depressive symptomatology. Minimum value = 0, maximum value = 15.

OTHER OUTCOMES:
Social Status Index and sociodemographical information | Baseline
  Hollingshead Index, age, sex, birth location
Cognitive reserve questionnaire | Baseline
  Cognitive reserve questionnaire (CRC), spanish version
Premorbid cognitive function | Baseline
  The Word Accentuation Test (TAP), spanish version

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Education, Psychology and Social Work; University of Lleida, Lleida
  - Cognitive disorders unity, Santa Maria's University Hospital, GSS, Lleida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calero García, M. D., & Navarro Gonzalez, E. (2006). Eficacia de un programa de entrenamiento en memoria en el mantenimiento de ancianos con y sin deterioro cognitivo. Clínica y Salud, 17(2), 187-202.
- [Background] Chang PJ, Wray L, Lin Y. Social relationships, leisure activity, and health in older adults. Health Psychol. 2014 Jun;33(6):516-23. doi: 10.1037/hea0000051. PMID 24884905
- [Background] Chiu HL, Chu H, Tsai JC, Liu D, Chen YR, Yang HL, Chou KR. The effect of cognitive-based training for the healthy older people: A meta-analysis of randomized controlled trials. PLoS One. 2017 May 1;12(5):e0176742. doi: 10.1371/journal.pone.0176742. eCollection 2017. PMID 28459873
- [Background] Dartigues JF, Foubert-Samier A, Le Goff M, Viltard M, Amieva H, Orgogozo JM, Barberger-Gateau P, Helmer C. Playing board games, cognitive decline and dementia: a French population-based cohort study. BMJ Open. 2013 Aug 29;3(8):e002998. doi: 10.1136/bmjopen-2013-002998. PMID 23988362
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755